CLINICAL TRIAL: NCT05006508
Title: Prevention and Development of Lifestyle Diseases With the Health and Lifestyle Tool
Brief Title: Prevention With the Health and Lifestyle Tool
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Lifestyle1
Record Dates: First submitted 2021-08-09; First posted 2021-08-16 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Intervention Model Description: Participants get access to the tool or get assigned to a control group without access.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usage of tool (Experimental): Participants get access to the tool and use it regularly
  Interventions: Behavioral: Lifestyle tool
- Controls on usual care (No Intervention): Participants who get randomized to control cannot access the tool and get no further follow-up. Their development of type 2 diabetes or development of HbA1c is tracked via clinical registries.

INTERVENTIONS:
Behavioral: Lifestyle tool — Regular use of the digital Lifestyle tool
  Arms: Usage of tool

SUMMARY:
In this study participants will be randomized to use a digital lifestyle tool over three years or to a control group without access to the tool. The investigators will prospectively via clinical registries follow the incidence and development of type 2 diabetes over three years in those using the tool regularly and those in the control group.

DETAILED DESCRIPTION:
Considerable evidence suggest that lifestyle changes can prevent or delay the onset of type 2 diabetes, and self-care behaviors largely determine HbA1c. Modifiable lifestyle factors have been established as key drivers of disease onset, progression, and prognosis, motivating the use of "lifestyle as medicine".

Digital health tools are increasingly incorporated into diabetes care, and have the potential to improve both behavioral and clinical outcomes on a broad basis. However, low levels of uptake, reduced user engagement over time, and low acceptance among patients, raise concerns about their effectiveness.

The objective or this study is to evaluate a new web-based tool, developed at the University Gothenburg, Sweden, that aims to support patient autonomy and motivation to make sustainable lifestyle changes.

The investigators will test the hypothesis that individuals who have access to the tool get lower incidence of type 2 diabetes or in case they already have diabetes develop improved glucose control compared with control individuals. The participants will complete the Findrisc questionnaire to assess the risk for type 2 diabetes to enable analysis of individuals with different risk.

The study is an investigator-initiated single-center study conducted over three years.

The tool is web-based and used via a computer or mobile phone. It is used at each individual's preferred pace but participants are recommended to login at least every other week. Every round the participants choose a themes (out of appr. 150 possible covering e.g. food, exercise, stress, self-reflection aspects), which takes appr. 15-30 minutes to complete. Participants then reflect on the content and how it could be implemented in daily life. When returning for next round participants are asked to reflect on any changes done since last time. There is no interaction between individual participants.

There will be two primary endpoints:

1. Incidence of type 2 diabetes as measured in non-diabetic participants with different risk for type 2 diabetes (controls vs. those using the tool regularly)
2. Change of HbA1c, reflecting long-term blood glucose control, from baseline to end of follow-up in participants who have type 2 diabetes (controls vs. those using the tool regularly).

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* Age above 35 years

Exclusion Criteria:

* type 1 diabetes, MODY or secondary diabetes
* conditions or treatments that in the judgement of the Investigator could affect the study evaluation
* connection with the study team, funders, authorities, universities or other public or private bodies in such a way that specific interests in the study outcomes could be suspected.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77000 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of type 2 diabetes | 3 years
  Incidence of type 2 diabetes defined as random plasma glucose >11.1 mmol/L or fasting glucose >7.0 mmol/L or HbA1C ≥6.5% compared between participants regularly using the tool and on usual care.
Change of long-term blood glucose concentration measured as glycated hemoglobin at end of follow-up | 3 years
  Intraindividual change of long-term blood glucose concentration measured as glycated hemoglobin (HbA1c) at end of follow-up relative to baseline compared between participants regularly using the tool and on usual care.
Prescription of anxiolytic medication | 3 years
  Number of participants on prescription of anxiolytic medication between participants regularly using the tool and on usual care.
Prescription of antidepessive medication | 3 years
  Number of participants on prescription of antidepressive medication between participants regularly using the tool and on usual care.

SECONDARY OUTCOMES:
Change of Anxiety estimated by General Anxiety Disorder 7-item scale | 1 year
  Change of Anxiety estimated by General Anxiety Disorder 7-item scale relative to baseline compared between participants regularly using the tool and on usual care. Score is from 0 to 21 with 21 meaning highest anxiety
Change of Patient Health Questionnaire 9-item scale | 1 year
  Change of Patient Health Questionnaire 9-item scale relative to baseline compared between participants regularly using the tool and on usual care. Score is from 0 to 27 with 27 meaning highest sign of depression

CONTACTS AND LOCATIONS:
Overall Officials: Anders Rosengren, Prof, Principal Investigator — Göteborg University
Locations (1):
- Anders Rosengrentest, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results will be shared after deidentification.
Time Frame: Data will be available after publication.
Access Criteria: To researchers who provide a methodologically sound proposal in order to achieve the aims of that proposal. Proposals should be directed by email to internetverktyg@gu.se

REFERENCES:
- [Derived] Dwibedi C, Abrahamsson B, Rosengren AH. Effect of Digital Lifestyle Management on Metabolic Control and Quality of Life in Patients with Well-Controlled Type 2 Diabetes. Diabetes Ther. 2022 Mar;13(3):423-439. doi: 10.1007/s13300-022-01214-2. Epub 2022 Feb 12. PMID 35150403